CLINICAL TRIAL: NCT06557408
Title: Factors Influencing the Occurrence of Pancreatic Fistula After Minimally Invasive Pancreatic Enucleation and Predictive Models: a Prospective Cohort Study
Brief Title: Pancreatic Fistula After Minimally Invasive Enucleation
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: CSPAC-MIEN-2
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Tumor, Benign; Pancreatic Neuroendocrine Tumor; Solid Pseudopapillary Tumor of the Pancreas
Keywords: Pancreatic benign or low-grade malignant tumors; Minimally invasive enucleation; Postoperative pancreatic fistula; Prediction model
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minimally invasive enucleation cohort: Surgical approaches to minimally invasive enucleation include laparoscopic or robotic-assisted procedures. During surgery, intraoperative ultrasonography is used to verify the position of the tumour in relation to the main pancreatic duct to ensure that injury to the main pancreatic duct is avoided and to help identify tumours within the pancreatic parenchyma. If injury to the main pancreatic duct is unavoidable, suture repair or bridging reconstruction techniques are used. If intraoperative freezing reveals the presence of high-grade dysplasia or invasive cancer, the procedure is converted to an oncological resection.

SUMMARY:
Patients suffering from postoperative pancreatic fistula (POPF) after minimally invasive enucleation (MIEN) show a characteristic pattern of longer duration and milder symptoms, which is different from pancreatic fistula after standard pancreatectomy. This study aimed to analyze the factors influencing clinically-relevant POPF (CR-POPF) after MIEN, investigate and develop a personalized predictive model for accurate prediction of CR-POPF.

DETAILED DESCRIPTION:
Minimally invasive enucleation (MIEN) has been widely used in managing benign and low-grade malignant pancreatic tumors, showing better protection of pancreatic function and better long-term outcomes compared to standard pancreatectomy.

However, the incidence of postoperative pancreatic fistula (POPF) after MIEN is higher compared to standard resection, mainly since a large part of the pancreatic wound is exposed, and the main pancreatic duct may be exposed or injured, etc. POPF is the most important postoperative complication, and it has become a major constraint to the conduct of pancreatic MIEN.

Although risk factors and predictive models for POPF in standard pancreatic surgery have been reported in the past, no predictive models have been reported specifically for MEN. With the increasing adoption of MIEN, there is an urgent need for a predictive model to guide the treatment and prognosis of POPF. Therefore, this study aims to conduct a cohort study, with data prospectively collected and retrospectively analyzed. The result of this study will provide a valuable reference for the development and application of MIEN.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years, regardless of gender.
2. Benign or low-grade malignant tumor of the pancreas.
3. Patients evaluated according to guidelines that indicate a need for surgery or a strong request for surgery.
4. Feasibility of performing minimally invasive pancreatic tumor enucleation based on preoperative imaging evaluation.
5. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Willingness to comply with the follow-up programme of the study and other protocol requirements.
7. Voluntary participation and signed informed consent.

Exclusion Criteria:

1. Concurrent presence of other malignant tumors.
2. Intraoperative frozen pathology or postoperative pathology indicating the tumor to be malignant, requiring oncological resection instead.
3. Severe impairment of cardiac, hepatic, or renal function (e.g., NYHA class 3-4 heart failure, ALT and/or AST levels exceeding three times the upper limit of normal, creatinine levels exceeding the upper limit of normal).
4. Missing data due to patient loss of followup, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of 182 consecutive patients who underwent MIEN at Fudan University Shanghai Cancer Center from July 2019 to November 2022. Nine patients with incomplete clinical data were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Clinically Relevant Postoperative Pancreatic Fistula | Within 90 days after surgery.
  Clinically Relevant Pancreatic Fistula including Grade B fistulas, which require treatment beyond simple drainage, as well as Grade C fistulas.

SECONDARY OUTCOMES:
Perioperative complication rate according to the Clavien-Dindo classification | Within 90 days after surgery.
  Adverse events occurring during or after surgery reported according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University; Xiaowu Xu, MD, Study Director — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center Shanghai, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crippa S, Bassi C, Salvia R, Falconi M, Butturini G, Pederzoli P. Enucleation of pancreatic neoplasms. Br J Surg. 2007 Oct;94(10):1254-9. doi: 10.1002/bjs.5833. PMID 17583892
- [Background] Zhou Y, Zhao M, Wu L, Ye F, Si X. Short- and long-term outcomes after enucleation of pancreatic tumors: An evidence-based assessment. Pancreatology. 2016 Nov-Dec;16(6):1092-1098. doi: 10.1016/j.pan.2016.07.006. Epub 2016 Jul 9. PMID 27423534
- [Background] Cauley CE, Pitt HA, Ziegler KM, Nakeeb A, Schmidt CM, Zyromski NJ, House MG, Lillemoe KD. Pancreatic enucleation: improved outcomes compared to resection. J Gastrointest Surg. 2012 Jul;16(7):1347-53. doi: 10.1007/s11605-012-1893-7. Epub 2012 Apr 24. PMID 22528577
- [Background] Giuliani T, De Pastena M, Paiella S, Marchegiani G, Landoni L, Festini M, Ramera M, Marinelli V, Casetti L, Esposito A, Bassi C, Salvia R. Pancreatic Enucleation Patients Share the Same Quality of Life as the General Population at Long-Term Follow-Up: A Propensity Score-Matched Analysis. Ann Surg. 2023 Mar 1;277(3):e609-e616. doi: 10.1097/SLA.0000000000004911. Epub 2021 Apr 14. PMID 33856383
- [Background] Duconseil P, Marchese U, Ewald J, Giovannini M, Mokart D, Delpero JR, Turrini O. A pancreatic zone at higher risk of fistula after enucleation. World J Surg Oncol. 2018 Aug 29;16(1):177. doi: 10.1186/s12957-018-1476-5. PMID 30157952
- [Background] Huttner FJ, Koessler-Ebs J, Hackert T, Ulrich A, Buchler MW, Diener MK. Meta-analysis of surgical outcome after enucleation versus standard resection for pancreatic neoplasms. Br J Surg. 2015 Aug;102(9):1026-36. doi: 10.1002/bjs.9819. Epub 2015 Jun 4. PMID 26041666
- [Background] Li Z, Zhuo Q, Shi Y, Chen H, Liu M, Liu W, Xu W, Chen C, Ji S, Yu X, Xu X. Minimally invasive enucleation of pancreatic tumors: The main pancreatic duct is no longer a restricted area. Heliyon. 2023 Nov 7;9(11):e21917. doi: 10.1016/j.heliyon.2023.e21917. eCollection 2023 Nov. PMID 38027678
- [Background] Liu R, Wakabayashi G, Palanivelu C, Tsung A, Yang K, Goh BKP, Chong CC, Kang CM, Peng C, Kakiashvili E, Han HS, Kim HJ, He J, Lee JH, Takaori K, Marino MV, Wang SN, Guo T, Hackert T, Huang TS, Anusak Y, Fong Y, Nagakawa Y, Shyr YM, Wu YM, Zhao Y. International consensus statement on robotic pancreatic surgery. Hepatobiliary Surg Nutr. 2019 Aug;8(4):345-360. doi: 10.21037/hbsn.2019.07.08. PMID 31489304
- [Background] Papachristou GI, Takahashi N, Chahal P, Sarr MG, Baron TH. Peroral endoscopic drainage/debridement of walled-off pancreatic necrosis. Ann Surg. 2007 Jun;245(6):943-51. doi: 10.1097/01.sla.0000254366.19366.69. PMID 17522520